CLINICAL TRIAL: NCT05451875
Title: Validation of Vital Signs Recording With VT-Patch® Connected Devices in Children
Brief Title: Validation of Vital Signs Recording With VT-Patch Connected Devices in Children
Acronym: VT
Status: Recruiting | Type: Observational
Sponsor: VitalTracer Ltd. (Industry)
Collaborators: St. Justine's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VT001
Record Dates: First submitted 2022-06-27; First posted 2022-07-11 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Vital Signs; Oxygen Saturation; Children; Intensive Care Unit; Heart Rate; Respiratory Rate
Keywords: Vital signs; SPO2; ECG; Continuous; Skin temperature; Heart rate; VitalTracer; Wearable; All-in-one; Children; PICU; Different Skin Color; Dark skin color; Monk Scale

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Non-invasive monitoring — Comparison of VitalTracer monitoring devices with invasive and/or non-invasive gold standard reference

SUMMARY:
: Patient readmission to PICU is a major point of concern for physicians because, although being a rare event, it has been strongly associated with more morbidity and death. Patient monitoring once they have left the PICU is drastically modified, and small connected devices could be an option to early identify patients at risk of PICU readmission. Such devices have been manufactured for the recording of vital signs in adults, but they do not exist for children.

Besides, studies have recently shown that devices that use optical sensors may be less accurate in individuals with dark skin pigmentation since dark skin tones impose a limitation on optical biometric sensing. The wearable and medical device industry has not sufficiently addressed this issue yet. This is one of the main challenges that need to be addressed in this area to make sure the connected devices using this technology will work with all different skin colours including very dark skin.

DETAILED DESCRIPTION:
Main objective: Assess the accuracy of VT-Patch® to measure oxygen saturation (SpO2) in children with diverse skin colour.

Secondary objectives: Assess the accuracy of VT-Patch® to measure 3 additional physiologic parameters (heart rate (HR), respiratory rate (RR), and temperature. Exploratory assessment of blood pressure (BP) measurement, ECG signal, and movement capture.

Design: Prospective validation study of VT-Patch® for the recording of 4 physiologic parameters and exploratory assessment of three additional parameters.

Methods: The study will be performed in two successive phases:

Run-in phase: Testing VT-Patch® on four children to assess the feasibility of the protocol.

Main study: validation phase of the devices on 12 children per age group (2 children per skin colour group) to assess its accuracy (VT-Patch® for less than 2 years old). The patients of the run-in phase will be included in the main study if no modification of the protocol is required. 5 physiologic parameters (HR, SpO2, RR, temperature, and ECG) will be prospectively and simultaneously recorded for 8 hours with VT-Patch® and the regular monitoring system implemented in the unit High-resolution database that will be the gold standard for evaluation. Vital signs recorded with the connected device will not be used for the clinical care of patients. The Skin colour of each patient will be assessed by the colorimetric Monk scale and as shown below.

ELIGIBILITY:
Inclusion Criteria:

* PICU monitoring for the next 24 hours

Exclusion Criteria:

* Recent cardiac or thoracic surgery
* Thoracic skin lesion that contraindicates the VT patch
* No parental consent
* Intermittent presence of one study observer in the patient room considered inappropriate by the physician or the nurse in charge because of the child's medical condition

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In order to achieve at least 80% match between physiological data's recorded with VT-Patch®, or VT-Watch® and with the standard of care (tolerated difference: 2% for SpO2), this study will include 10 patients per age group (see below) including 4 patients per age group with invasive arterial pressure monitoring (arterial line).
  1. Neonates: 0 - 28 days
  2. Infants:29 days - 2 years
  3. Children: 2 - 12 years
  4. Adolescents:12 - 18 years
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of VitalTracer devices Oxygen Saturation (SPO2) measurement for different skin colour | 8 hours per subject
  Percentage of the difference between the absolute value of SpO2 recorded by VT-Patch and the one recorded in high resolution database.

SECONDARY OUTCOMES:
Accuracy of VitalTracer devices blood pressure, heart rate, skin temperature, and Electrocardiogram (ECG) measurement | 8 hours per subject
  Percentage of the difference between the absolute value of Blood Pressure, Heart Rate and skin temperature and the quality of ECG signals recorded by the VT-Patch and the one recorded in high resolution database.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte Justin Hospital, Montreal, Quebec, Canada